CLINICAL TRIAL: NCT07395934
Title: Comparison of Continuous Epidural Infusion vs. Programmed Intermittent Epidural Bolus Combined With Patient-Controlled Epidural Analgesia for Labor Pain Relief: A Randomized Controlled Trial
Brief Title: Comparing PIEB and CEI for Labor Pain Relief
Acronym: COPILOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Da Nang Family General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/2025/BVGD-HDĐĐ
Record Dates: First submitted 2026-01-18; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Labor Pain; Analgesia, Epidural; Analgesia, Obstetrical; Labor, Obstetric
Keywords: Programmed Intermittent Epidural Bolus (PIEB); Continuous Epidural Infusion (CEI); Patient-Controlled Epidural Analgesia (PCEA); Visual Analog Scale (VAS)
MeSH Terms: conditions — Labor Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIEB Group (Experimental): Maintenance of labor analgesia using Programmed Intermittent Epidural Bolus.
  Interventions: Procedure: PIEB + PCEA
- CEI Group (Active Comparator): Maintenance of labor analgesia using Continuous Epidural Infusion.
  Interventions: Procedure: CEI + PCEA

INTERVENTIONS:
Procedure: PIEB + PCEA — Initial dose: 10 mL (0.1% Ropivacaine + 2 mcg/mL Fentanyl). Maintenance: 8 mL bolus every 60 mins. PCEA: 5 mL bolus, 10-min lockout.
  Arms: PIEB Group
Procedure: CEI + PCEA — Initial dose: 10 mL (0.1% Ropivacaine + 2 mcg/mL Fentanyl). Maintenance: Continuous infusion at 8 mL/hour. PCEA: 5 mL bolus, 10-min lockout.
  Arms: CEI Group

SUMMARY:
The purpose of this randomized controlled trial is to compare the efficacy and safety of two epidural analgesia maintenance methods for labor pain relief: Programmed Intermittent Epidural Bolus (PIEB) and Continuous Epidural Infusion (CEI), both combined with Patient-Controlled Epidural Analgesia (PCEA). The study aims to evaluate which technique provides superior analgesia while minimizing anesthetic consumption and preserving maternal motor function. A total of 60 parturients at Family Hospital, Da Nang, will be randomly assigned to either the PIEB or CEI group. Outcomes including pain intensity (VAS scores), total drug consumption, maternal satisfaction, and neonatal Apgar scores will be assessed.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial conducted at the Labor and Delivery Unit of Family Hospital, Da Nang. The investigation focuses on the clinical advantages of automated high-pressure bolus delivery (PIEB) compared to constant low-pressure flow (CEI) in optimizing the spread of local anesthetics within the epidural space.

Clinical Procedures: All participants receive a standardized initial manual bolus of 10 mL (0.1% Ropivacaine and 2 mcg/mL Fentanyl) to establish a baseline sensory block. Following this induction, patients are managed according to their assigned study arm:

PIEB Group: Analgesia is maintained using a programmed pump set to deliver an automated bolus of 8 mL every 60 minutes, starting one hour after the initial dose.

CEI Group: Analgesia is maintained via a continuous infusion of the same anesthetic solution at a constant rate of 8 mL/hour.

Analgesia Management and Rescue Protocol: Both groups have access to PCEA, allowing for self-administered 5 mL boluses with a 10-minute lockout period, capped at a maximum of 20 mL per hour.

To ensure maternal comfort, a standardized rescue protocol is strictly followed: if the Visual Analog Scale (VAS) score remains > 4 after two consecutive PCEA demands, a manual rescue bolus of 5 mL is administered by the anesthesia team.

ELIGIBILITY:
Inclusion Criteria:

* Parturients indicated for labor analgesia for vaginal delivery via epidural anesthesia.
* Age from 18 to 40 years.
* Physical status: ASA II.
* Singleton pregnancy, full-term, vertex presentation in labor.
* Indication for vaginal delivery.
* No contraindications to epidural anesthesia.
* Agreement to participate in the research and signed written informed consent.

Exclusion Criteria:

* Contraindications to epidural analgesia.
* History of allergy to local anesthetics (Ropivacaine) or opioids (Fentanyl).
* High-risk pregnancies: Preeclampsia, placenta previa, placental abruption.
* Fetal distress or fetal abnormalities.
* Chronic use of analgesic drugs or neurological/psychiatric disorders.
* Parturients who refuse to participate or request to withdraw from the research.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Labor Pain Intensity | Baseline (prior to epidural analgesia induction), then at 5 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours after the initiation of analgesia. Additional assessments are performed at full cervical dilation, during the fetal expulsion stage
  Pain intensity is assessed using the Visual Analog Scale (VAS), a self-reported scale where 0 represents "no pain" and 10 represents "the worst pain imaginable". Lower scores indicate better analgesic efficacy. Score on a scale from 0 to 10.

SECONDARY OUTCOMES:
Total Ropivacaine Consumption | From the initiation of epidural analgesia until the completion of perineal repair, assessed up to 24 hours.
  The total dose of Ropivacaine (in milligrams) administered to each participant throughout the entire labor and delivery process. This sum includes the 10 mg initial manual bolus , the programmed intermittent boluses (8 mg/hour) or continuous infusion (8 mg/hour) , and any 5 mg patient-controlled epidural analgesia (PCEA) or manual rescue doses administered.
Incidence of Maternal Motor Block | From the initiation of epidural analgesia, assessed at 5, 10, 30, 60 minutes, then every 2 hours until the completion of perineal repair (assessed up to 24 hours).
  The presence and severity of motor blockade are evaluated using the Modified Bromage Scale (0 = No motor block; 1 = Inability to raise extended legs; 2 = Inability to flex knees; 3 = Inability to flex ankles). Higher scores mean a worse outcome (greater motor impairment).
Maternal Satisfaction Score | At 2 hours after the completion of perineal repair (assessed up to 24 hours after enrollment).
  Overall satisfaction is assessed using a 5-point Likert scale. The scale ranges from 1 to 5, where 1 indicates "Not Satisfied" and 5 indicates "Very Satisfied". Higher scores mean a better outcome (greater satisfaction).
Neonatal Apgar Scores | At 1 minute and 5 minutes post-delivery.
  Newborn health is assessed using the Apgar Scale. The total score ranges from 0 to 10, calculated based on five criteria (each scored 0-2). Higher scores mean a better outcome (better neonatal condition).

CONTACTS AND LOCATIONS:
Locations (1):
- Family General Hospital, Da Nang, Vietnam